CLINICAL TRIAL: NCT06706219
Title: Efficacy and Safety of Sacituzumab Tirumotecan (SKB264) in Combination With Pembrolizumab in Patients With Initially Unresectable Stage III Non-small Cell Lung Cancer (NSCLC): a Multi-center Phase II Study
Brief Title: Efficacy and Safety of SKB264 in Combination With Pembrolizumab in Patients With Initially Unresectable Stage III NSCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Director, Head of Medical Oncology, Principal Investigator, Clinical Professor, Hunan Province Tumor Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeoTrop
Record Dates: First submitted 2024-11-23; First posted 2024-11-26 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Non Small Cell Lung Cancer (Stage III)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sacituzumab tirumotecan (SKB264) in combination with pembrolizumab (Experimental)
  Interventions: Drug: Sacituzumab tirumotecan plus pembrolizumab

INTERVENTIONS:
Drug: Sacituzumab tirumotecan plus pembrolizumab — Participants meeting the inclusion criteria will receive pembrolizumab 200 mg IV on D1, Q3W + SKB264 4mg/kg IV on D1, D15 and D29，Q2W for 12 weeks as induction therapy.
  Subjects who receive radical radiotherapy will undergo 8 cycles of pembrolizumab 200 mg IV on D1, Q3W; For those receiving surgical treatment, pembrolizumab is selected for adjuvant therapy for pCR patients, and SKB264 combination with pembrolizumab is selected non-PCR patients.

SUMMARY:
This study is a phase 2 open-label, multicenter clinical study to evaluate the efficacy and safety SKB264 in combination with pembrolizumab in patients with unresectable stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
This study is a phase 2 open-label, multicenter clinical study to evaluate the efficacy and safety SKB264 in combination with pembrolizumab in patients with unresectable stage III non-small cell lung cancer. The study includes a screening period (up to 28 days after the subject signs the informed consent form until before the first dose), a treatment period (including an induction treatment period, a local treatment period (surgery or radical radiotherapy), and a consolidation treatment period), and a follow-up period (including two parts of safety follow-up and survival follow-up).

Approximately 50 patients with initially unresectable stage III non-small cell lung cancer patients, without EGFR/ALK/ROS-1-sensitive mutations, without chest radiotherapy and systemic anti-tumor therapy, were enrolled and treated with Sacituzumab tirumotecan (SKB264) in combination with pembrolizumab until disease progression, intolerable toxicity, or meeting the criteria for discontinuation of the trial drug.

The primary endpoint is the investigator-assessed 18-month progression-free survival (PFS) rate of intention-to-treat population (ITT). Secondary endpoints include event-free survival (EFS), overall survival (OS), R0 surgical resection rate, complete response (pCR) rate, major pathological response (MPR) rate and safety, objective response rate (ORR) in the induce treatment period. Recruitment for the study is expected to begin in mainland China around January 2025, with the trial anticipated to conclude in January 2028.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients who voluntarily participate in this clinical study, understand the study procedures and are able to sign the informed consent form in writing;
* 2.Men or women aged 18-70 years (inclusive) at the time of signing the informed consent form.
* 3.ECOG PS score of 0 or 1.
* 4.Histologically or cytologically confirmed stage III squamous cell or non-squamous cell non-small cell lung cancer that cannot be surgically treated as determined by the investigator. Disease staging should be based on the American Joint Committee on Cancer (AJCC)/Union for International Cancer Control (UICC) NSCLC staging system, 8th edition.
* 5.Ability to provide tumor tissue specimens, either archived within 6 months prior to the first dose of study drug or freshly obtained. See the laboratory manual for specific requirements.
* 6.Pulmonary function of at least FEV1 > 1.0 L and FEV1% > 40% within 3 months.
* 7.Patients must have measurable target lesions examined by CT or MRI per RECIST v1.1 criteria. Tumor imaging assessments are performed within 28 days prior to the first dose.
* 8.Adequate hematologic and vital organ functions, as defined by the following laboratory findings, which need to be completed within 14 days prior to the first study treatment:

  1. Hematology (no hematopoietic stimulating factor drugs or blood transfusion within 14 days before the first study treatment): absolute neutrophil count (ANC) ≥ 1.5 × 109/L, absolute lymphocyte count (LC) ≥ 0.5 × 109/L; platelet count (PLT) ≥ 100 × 109/L, hemoglobin (Hb) ≥ 90 g/L
  2. Liver function: aspartate transferase (AST) and alanine aminotransferase (ALT) ≤2.5 x ULN; ; serum total bilirubin (TBIL) ≤ 1.5 x ULN (total bilirubin ≤ 3.0 mg/dL in patients with confirmed Gilbert syndrome); albumin (ALB) ≥ 3 g/dL;
  3. Renal function: creatinine clearance rate (CrCl) ≥ 45 mL/minute (by Cockcroft-Gault formula);
  4. Coagulation: international normalized ratio (INR) ≤ 1.5, activated partial thromboplastin time (APTT) ≤ 1.5 x ULN;
  5. Cardiac color ultrasound: left ventricular ejection fraction (LVEF) ≥ 50%
* 9.Female patients of childbearing potential must have a negative pregnancy test (serum or urine) within 72 hours prior to receiving the study drug. Reliable contraception, such as intrauterine devices, oral contraceptives, or condoms, must be used during the trial and for 90 days following the final dose. Male participants with partners of childbearing potential must use condoms during the trial and for 30 days following the studys conclusion

Exclusion Criteria:

* 1.Histologically or cytologically confirmed mixed SCLC and NSCLC, large cell neuroendocrine carcinoma and sarcomatoid carcinoma;
* 2.Patients with positive EGFR mutations or ALK gene rearrangements. All patients must undergo EGFR gene testing and ALK gene and/or immunohistochemistry testing；
* 3.Presence of malignant pleural effusion. If a patient has a extractable pleural effusion during the screening period, at least one thoracentesis must be performed to confirm whether there are malignant tumor cells;
* 4.Patients who have received any systemic anti-tumor therapy for NSCLC, including surgical treatment, local radiotherapy, cytotoxic drug therapy, targeted therapy, immunotherapy, or traditional Chinese medicine (excluding patients who had other malignancies that were radically resected and have remained recurrence-free for more than 5 years);
* 5.Diagnosis of any other cancer within 5 years prior to enrollment, except for carcinoma in situ of the cervix, cured basal cell carcinoma, or bladder epithelial tumors (including Ta and Tis);
* 6.Patients with active autoimmune diseases or a history of autoimmune conditions, such as uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, or hypothyroidism (the latter is allowed if controlled by hormone replacement therapy), or tuberculosis. Note: Patients with a history of childhood asthma that has completely resolved and has not required treatment in adulthood may be included. Patients with skin conditions (e.g., vitiligo, psoriasis, or alopecia) that do not require systemic therapy are also eligible;
* 7.Patients with current or prior history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-induced pneumonitis, radiologically confirmed active pneumonitis, or severe pulmonary impairment;
* 8.Patients who have received systemic corticosteroids (prednisone >10 mg/day or equivalent) or other immunosuppressive medications within 2 weeks prior to the first dose. Inhaled or topical corticosteroids and adrenal replacement therapy are allowed if there is no evidence of active autoimmune disease, and the dose of prednisone is less than 10 mg/day;
* 9.Known hypersensitivity to the investigational drug or any of its components;
* 10.Patients who are active carriers of hepatitis B, hepatitis C, or HIV;
* 11.Pregnant or breastfeeding women;
* 12.Patients of childbearing potential who are unwilling or unable to use effective contraception. Additionally, patients with a history of neurological or psychiatric disorders who demonstrate poor treatment compliance;
* 13. Any other condition that, in the investigator's opinion, makes the patient unsuitable for participation in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
18m EFS rate | Time from the first dose treatment to 18 months
  18-month progression-free survival (PFS) rate

SECONDARY OUTCOMES:
Event-free survival (EFS) | Time from first subject enrollment to study completion, or up to 60 months
  Defined as the time from the first dose treatment to the occurrence of any event, including disease progression, discontinuation of treatment for any reason, or death.
R0 surgical resection rate | Time from the first subject dose to study completion, or up to 60 months
  No residual ratio under the microscope after surgical resection
Complete Response (pCR) rate | Time from the first subject dose to study completion, or up to 60 months
  Defined as the absence of active tumors in lesions at the time of surgical resection of primary tumors.
Major Pathological Response (MPR) rate | Time from the first subject dose to study completion, or up to 60 months
  Defined as the incidence of ≤10% active tumors in lesions at the time of surgical resection of primary tumors.
Objective response rate (ORR) | Time from the first subject dose to study completion, or up to 60 months
  The ORR of ITT after SKB264 combined with pembrolizumab was evaluated according to the investigator's Solid Tumor Response Assessment Criteria (RECIST) version 1.1, defined as the proportion of subjects who were evaluated for complete response (CR) + partial response (PR) after induce treatment
Adverse events (AEs) | From the first dose to 28 days after the last dose, until 36 months
  Number of participants with adverse events (AEs) according to CTCAE 5.0
Overall survival (OS) | Time from the first subject dose to study completion, or up to 60 months
  Defined as the time from the first dose treatment to death.

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Provincal Tumor Hospital, Changsha, Hunan, China